CLINICAL TRIAL: NCT04629066
Title: Efficacy and Safety of ICD Remote Monitored Exercise Testing to Improve Heart Failure Outcomes: REMOTE HF-ACTION (Pilot Randomized Controlled Trial)
Brief Title: Efficacy and Safety of ICD Remote Monitored Exercise Testing to Improve Heart Failure Outcomes: REMOTE HF-ACTION
Acronym: x
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Evaluation System for health Technology Coordinating Center (Other); Medical Device Innovation Consortium (MDIC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00107053
Record Dates: First submitted 2020-11-02; First posted 2020-11-16 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure
Keywords: Remote Exercise Prescription; Cardiac Implant
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Usual care will include regularly scheduled visits with the clinical heart failure care team and medical therapy as prescribed by that team.
- Remote prescription for aerobic exercise (Experimental): The exercise prescription will be created by an exercise physiologist after incorporating remotely collected data from a patient directed smartphone app assessing HF symptom severity, vital signs, weight, and blood sugar, and cardiac implant measures of physical activity, heart rate, heart failure volume status and heart rhythm, and Fitbit measures of physical activity.
  Interventions: Behavioral: Remote Cardiac Rehabilitation (CR)

INTERVENTIONS:
Behavioral: Remote Cardiac Rehabilitation (CR) — Patients randomized to remote CR will be asked to use an app for cardiac rehabilitation a minimum of 3 times a week. Patients will be given an exercise prescription provided by a certified exercise physiologist.
  The exercise prescription will change each week based on refreshed data from the prior week.
  Instructional videos for each exercise are provided in the app. Patients will not be told to perform the exercise at a particular time. Instead they will be asked to complete a certain amount of exercise per week at whatever time is convenient for them. Patients randomized to remote CR will also receive App based reminders to take their medications, resources to guide healthy eating habits, and other behavioral health advice as is done as standard of care in both remote based and clinic based CR.
  Arms: Remote prescription for aerobic exercise

SUMMARY:
This single center randomized controlled trial will involve 50 medically stable outpatients with HF, reduced ejection fraction, and previously implanted ICD or CRT-D devices followed longitudinally on the Abbott Medical Merlin remote patient monitoring network. Patients will be randomized in a 1:1 fashion to usual care plus a remotely administered home based weekly prescription for aerobic exercise (intervention) or usual care alone (control). Usual care will include regularly scheduled visits with the clinical heart failure care team and medical therapy as prescribed by that team. The exercise prescription will be created by an exercise physiologist after incorporating remotely collected data from a patient directed smartphone app assessing HF symptom severity, vital signs, weight, and blood sugar, implantable device measures of physical activity, heart rate, heart failure volume status and heart rhythm, and Fitbit measures of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients have a MERLIN patient registry record for an ICD or CRT-D implantation between 01/01/2010-12/31/2020
* Age > 18 years
* Left ventricular ejection fraction < 50% by echocardiogram, nuclear cardiology scan, cardiac magnetic resonance imaging, or invasive left ventriculography within the past 12 months.
* Ongoing NYHA class II, III, or IV HF symptoms by questionnaire
* Ongoing use of beta-blocker and ACE-inhibitor or angiotensin receptor blocker or willingness to start them- assessed by Duke Epic EMR screening.
* Life expectancy > 12 months
* To allow for a post-surgical adjustment period, patients must be >30 days out from device implantation

Exclusion Criteria:

* Prior participation in CR- by patient questionnaire
* Unwillingness to sign informed consent form
* Currently performing > 240 minutes of device detected daily PA- by ICD/CRTD remotely collected data.
* Lack of a smartphone or unwillingness to use an App or Fitbit device
* Prior left ventricular assist device (LVAD) implantation or heart transplantation
* ICD tachyarrhythmia therapies programmed off
* Inherited arrhythmia condition with contraindication to exercise (eg Lamin A mutation or ARVC)
* No transmissions through Merlin.net in past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Atwater, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Remote Prescription for Aerobic Exercise: The exercise prescription will be created by an exercise physiologist after incorporating remotely collected data from a patient directed smartphone app assessing HF symptom severity, vital signs, weight, and blood sugar, and cardiac implant measures of physical activity, heart rate, heart failure volume status and heart rhythm, and Fitbit measures of physical activity.
  Remote Cardiac Rehabilitation (CR): Patients randomized to remote CR will be asked to use an app for cardiac rehabilitation a minimum of 3 times a week. Patients will be given an exercise prescription provided by a certified exercise physiologist.
  The exercise prescription will change each week based on refreshed data from the prior week.
  Instructional videos for each exercise are provided in the app. Patients will not be told to perform the exercise at a particular time. Instead they will be asked to complete a certain amount of exercise per week at whatever time is convenient for them. Patients randomized to remote CR will also receive App based reminders to take their medications, resources to guide healthy eating habits, and other behavioral health advice as is done as standard of care in both remote based and clinic based CR.
Period: Overall Study
Arm/Group | Usual Care | Remote Prescription for Aerobic Exercise
Started | 7 | 6
Completed | 4 | 4
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Remote Prescription for Aerobic Exercise | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.89) | 58.8 (10.46) | 63.8 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Abbott Implantable Cardioverter-defibrillator (ICD) or Cardiac Resynchronization Therapy Defibrillator (CRT-D) Device Measured Daily Physical Activity (PA)
Description: Reported in minutes of PA per day.
Time Frame: 12 weeks after randomization
Population: Data not collected on two participants.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Usual Care | Remote Prescription for Aerobic Exercise
Number analyzed (Participants) | 5 | 6
minutes per day | 129.3 (77.96) | 171.4 (74.59)

2. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Heart Failure (HF) Symptoms Severity Score
Description: The KCCQ has a range of 0 to 100, where a higher score indicates a more favorable health status.
Time Frame: Baseline to 12 weeks
Population: Data not collected on six participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Remote Prescription for Aerobic Exercise
Number analyzed (Participants) | 3 | 2
score on a scale | 5.2 (9.02) | 11.5 (16.20)

3. Secondary Outcome: Number of Heart Failure Hospitalization, Fracture, Myocardial Infarction, Serious Adverse Arrhythmia, and ICD Therapy Combination Events
Time Frame: Cumulative during 12 weeks of intervention
Measure: Number; unit: events
Arm/Group | Usual Care | Remote Prescription for Aerobic Exercise
Number analyzed (Participants) | 7 | 6
events | 1 | 1

4. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Heart Failure (HF) Symptom Severity Score
Description: The KCCQ has a range of 0 to 100, where a higher score indicates a more favorable health status.
Time Frame: 12 weeks after randomization
Population: Data not collected on six participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Remote Prescription for Aerobic Exercise
Number analyzed (Participants) | 3 | 2
score on a scale | 86.1 (14.63) | 93.8 (8.84)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected between consent and study completion, for a total of 13 weeks.
Arm/Group | Usual Care | Remote Prescription for Aerobic Exercise
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=7) | Remote Prescription for Aerobic Exercise (N=6)
Stent Placement (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=7) | Remote Prescription for Aerobic Exercise (N=6)
Back injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT04629066/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT04629066/SAP_001.pdf